CLINICAL TRIAL: NCT02812407
Title: Baseline Impedance Measured on High Resolution Esophageal Impedance Manometry to Discriminate GERD From Non GERD Patients
Brief Title: HRIM vs Mucosal Impedance in GERD Participants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No linger a clinically relevant research question
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karthik Ravi, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-003580
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2019-09

CONDITIONS: Gastro-esophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mucosal Impedance (Experimental): Patient's having a clinically indicated endoscopy, a high resolution impedance manometry and a 24 hour pH impedance study.
  During the clinical endoscopy, the 2.13 mm catheter will be passed through the channel of the standard endoscope this is called an Intraluminal Impedance. This device has not been approved by the Food and Drug Administration (FDA) but it is considered to be minimal risk related to using it.
  Interventions: Device: Mucosal Impedance

INTERVENTIONS:
Device: Mucosal Impedance — During the clinical endoscopy, the 2.13 mm catheter will be passed through the channel of the standard endoscope this is called an Intraluminal Impedance. The Intraluminal impedance (made by Sandhill Scientific) has not been approved by the Food and Drug Administration (FDA) but it is considered to be minimal risk related to using it. The catheter gives the investigators a reading at each level.
  * The catheter will be placed on the esophageal mucosa 5 cm above the gastroesophageal junction (where the stomach and esophagus meet) for 5 second
  * At 10 cm above the gastroesophageal junction the catheter will be placed for 5 seconds
  * And at 20 cm
  Other Names: Impedance

SUMMARY:
Does baseline impedance measured during the landmark phase of esophageal High resolution impedance manometry HRIM correlates with direct mucosal impedance measurement and discriminates GERD from non GERD patients?

DETAILED DESCRIPTION:
Patients referred to the Mayo Clinic Rochester for a clinically indicated high resolution impedance manometry (HRIM), 24 hour impedance pH (MII-pH) study, and esophagogastroduodenoscopy (EGD) will be recruited. Gastroesophageal reflux will be defined as a total 24 hour esophageal acid exposure time ≥5% regardless of concomitant Proton Pump inhibitor (PPI) use. A negative 24 hour MII-pH study will be defined as an acid exposure time ≤2% off PPI therapy or ≤1% if on PPI therapy.

ELIGIBILITY:
Patients being seen at Mayo clinic Rochester having a clinically indicated endoscopy, a high resolution impedance manometry and a 24 hour pH impedance study.

Inclusion criteria:

* Adults ages 18-90
* Patients scheduled for or have completed a HRIM ( within 5 days)
* Patients scheduled for or recently have completed a MII-pH studies ( within 5 days)
* Patients scheduled for EGD

Exclusion criteria:

* Technically limited esophageal HRIM or MII-pH study
* Patients with HRIM and MII-pH studies not performed within 5 days of each other
* Patients with EGD not performed within 30 days of HRIM and MII-pH studies
* Medical conditions such as severe heart or lung disease that preclude safe performance of endoscopy
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
The mean impedance | 2 years
  The mean impedance measured in Ohms as a measure of mucosal integrity and surrogate for GERD

SECONDARY OUTCOMES:
Maximal impedance measured on HRIM in GERD patients compared to minimal impedance in patients without GERD to determine a potential diagnostic cutoff value | 2 years
  Evaluate the measurement of HRIM and mucosal impedance in patients that did not show gastroesophageal reflux disease per the HRIM and impedance testing

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ravi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials